CLINICAL TRIAL: NCT03178448
Title: PolyvasculaR Evaluation for Cognitive Impairment and vaScular Events (PRECISE)
Brief Title: PolyvasculaR Evaluation for Cognitive Impairment and vaScular Events
Acronym: PRECISE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, Professor, Beijing Tiantan Hospital
Other Study IDs: 2016YFC0901001
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples will also be collected at baseline to test genetic and metabolomic markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to characterize the prevalence of clinical or subclinical polyvascular lesions and 4-year progression rate of plaque in intracranial and carotidal arteries in a Chinese community population using vascular imaging techniques; to investigate the both traditional and emerging genetic, metabolomic, and environmental risk factors of presence and progression of intracranial and carotidal plaque; and to investigate the association between polyvascular lesions and future risk of cognitive impairment, cardio-/cerebrovascular events and death.

DETAILED DESCRIPTION:
Atherosclerosis is the most common cardiovascular disease and accounts for the greatest number of cardiovascular and cerebrovascular events and death. Polyvascular lesions with coexistent lesions (especially atherosclerosis) in multiple arterial territories (at least 2 of coronary, cerebral, lower extremity arteries), could be associated with higher risk of future cardio-/cerebrovascular diseases. However, previous studies either roughly defined polyvascular diseases according to established clinically recognized arterial diseases in multiple arterial territories, or tested multiterritorial subclinical atherosclerosis without tests of intracranial and peripheral arteries. Furthermore, recent research also showed that cardiometabolic diseases and cardiovascular risk factors are associated with worse cognitive abilities. A thorough evaluation of multiterritorial lesions in whole body used advanced vascular imaging techniques is required to precisely assess the association of polyvascular lesions with future cardio-/cerebrovascular events and cognitive impairment.

Additionally, Asian population might have higher prevalence of intracranial atherosclerosis than the Caucasian, and intracranial atherosclerosis is the most common cause of ischemic stroke in Asia population. However, there are limited data about the prevalence and progression of intracranial atherosclerosis in Chinese population. More and more studies have shown that presence and progression of atherosclerotic plaque is not only related to the degree of stenosis, but also with plaque characteristics such as rich lipid core, plaque hemorrhage and inflammatory cell infiltration. High-resolution magnetic resonance (HR-MRI) can not only show the degree of arterial stenosis, the size of atherosclerotic plaque, but also can analyze the composition of the plaque to assess the stability of the plaque. HR-MRI techniques enable early detection of atherosclerosis, characterization of the atherosclerotic composition and burden. It is important to estimate the prevalence and progression rate of intracranial atherosclerotic plaque based on HR-MRI and to estimate its traditional and emerging determinants in Chinese population.

In this study, a total of 3000 subjects aged 50 to 75 years from 6 villages and 4 communities in Lishui city, Zhejiang province, China, will be enrolled. All the eligible subjects in the selected villages/community will be enrolled based on cluster sampling.

All the participants will be interviewed at baseline and followed up for 4 years. Data collection at baseline will be performed through face-to-face interviews by trained interviewers (neurologists from participating hospitals) with a standardized protocol. Baseline data include demographics, medical history, cardiovascular risk factors, dietary habits, physical activity, lifestyle, medication use, electrocardiogram, vascular imaging tests and Montreal Cognitive Assessment (MoCA). Blood and urine samples will also be collected at baseline to test genetic and metabolomic markers.

The sequences of brain MRI included T1,T2, FLAIR, DWI,ADC,MRA,SWI,T2*,T1-VISTA, SNAP,3D-T1,resting-state fMRI and DTI. Baseline vascular imaging tests include HR-MRI sequences in intracranial and carotidal arteries, computed tomographic angiography (CTA) in coronary, aorta, renal, hepatic, pancreatic and iliofemoral arteries, and fundus fluorescein photography (retinal photography) in retinal vessel. All MRI scans were performed on 3.0 T Philips scanners. CTA scans were performed on third-generation dual-source Siemens system (SOMATOM Force). HR-MRI sequences were performed both at baseline and after 4 years to identify intracranial and carotidal atherosclerotic stenosis and plaque and measure the intracranial and carotidal vessel wall, lumen area, and plaque when present. Additionally, heart function will be tested using color Doppler echocardiography, and ankle-brachial index will be tested using Doppler ultrasound. All the imaging techniques will be conducted in a fixed machine by fixed trained investigators based on a standardized protocol. These imaging techniques enable early detection of intracranial and extracranial vascular lesions, characterization of the atherosclerotic composition and burden, and monitoring of plaque progression in intracranial and carotidal arteries.

Routine follow-up will be performed each year to collect cardio-/cerebrovascular events and death after enrollment. A further face-to-face interview will be performed at 2 years and 4 years to collect brain MRI scanning and cognitive impairment. At 2-year and 4-year follow-up visits, standard clinical and neuropsychologic assessments will be performed, including MoCA, Mini-Mental State Exam scores, Geriatric Depression Scale, Digit Span, Rey Auditory Verbal Learning Test, Rey-Osterrieth Complex Figure Test, Trail Making A and B, Stroop Task, Verbal Fluency Test, Boston Naming Test, Clock Drawing Test, Symbol Digit Modalities Test, Neuropsychiatric Inventory and Clinical Dementia Rating. Fasting blood and morning urine samples will be collected at each follow-up visit following same protocol as that at baseline.

The protocol of this study was approved by the ethics committee of Beijing Tiantan Hospital and Lishui Hospital of Zhejiang University. All participants provided written informed consents before entering the study.

ELIGIBILITY:
Inclusion Criteria:

* Community population in Lishui city;
* Age between 50 and 75 years.

Exclusion Criteria:

* Mental illness;
* Advanced cancers or any disease that decreases life expectation to ≤4 years;
* Allergy to iodine contrast, renal failure with creatinine clearance <60 mL/min, or blood urea nitrogen (BUN) or creatinine (CR) more than upper limit of the normal range that contraindicates CTA;
* Pacemaker, implantable automatic defibrillator, or any implanted device that contraindicates MRI.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population of the study consists of community population aged 50-75 years in Lishui city in southeast of China.
Sampling Method: Probability Sample
Enrollment: 3067 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
New composite vascular event 1 | 4 years
  Any new event of nonfatal stroke (ischemic or hemorrhagic), nonfatal myocardial infarction (MI) or cardiovascular death (including fatal stroke, fatal MI, and other cardiovascular death).
New composite vascular event 2 | 4 years
  Any new event of nonfatal stroke, nonfatal MI, cardiovascular death, vascular interventions (bypass graft, angioplasty, stent and amputation for ischemia), or hospitalizations for vascular events (including unstable angina pectoris, transient ischemic attack (TIA) and other ischemic arterial event including worsening of peripheral vascular disease (PAD)).

SECONDARY OUTCOMES:
Prevalence of polyvascular lesions, including atherosclerotic stenosis and plaque; | at baseline
4-year progression rate of atherosclerotic plaque in intracranial and carotidal arteries. | 4 years
Fatal or nonfatal MI; | 4 years
Fatal or nonfatal stroke; | 4 years
Transient ischemic attack (TIA) | 4 years
All causes of death (cardiovascular or noncardiovascular death); | 4 years
Hospitalizations for vascular events; | 4 years
Vascular interventions; | 4 years
  Vascular interventions such as arterial bypass, balloon dilatation, stent implantation, carotid endarterectomy, mechanical thrombolysis and ischemic amputation.These events will be collected by self-reported by participants and confirmed by reviewing their medical records.
Other vascular events (PAD, subclavian steal syndrome and systemic thromboembolic events); | 4 years
New diagnosed diabetes mellitus; | 4 years
New diagnosed chronic kidney disease; | 4 years
Cognitive impairment measured by the Montreal Cognitive Assessment (MoCA). | 4 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Lishui Hospital of Zhejiang University (the Central Hospital of Lishui), Lishui, Zhejiang
  - Beijing Tiantan Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
The data can be requested through the website of the data management system (http://paper.ncrcnd.org.cn/) or by sending email to the principal investigators.

REFERENCES:
- [Derived] Zhou M, Mei L, Jing J, Yang Y, Cai X, Meng X, Jin A, Lin J, Li S, Li H, Wei T, Wang Y, Wang Y, Pan Y. Blood Pressure Partially Mediated the Association of Insulin Resistance and Cerebral Small Vessel Disease: A Community-Based Study. J Am Heart Assoc. 2024 Mar 5;13(5):e031723. doi: 10.1161/JAHA.123.031723. Epub 2024 Feb 23. PMID 38390815
- [Derived] Cai X, Sun J, Jin A, Jing J, Wang S, Mei L, Meng X, Li S, Wei T, Wang Y, Pan Y. Association of insulin resistance with intra- and extra-cranial atherosclerotic burden in the nondiabetic community population. Neurobiol Dis. 2023 Oct 1;186:106268. doi: 10.1016/j.nbd.2023.106268. Epub 2023 Aug 23. PMID 37625526
- [Derived] Tian Y, Cai X, Zhou Y, Jin A, Wang S, Yang Y, Mei L, Jing J, Li S, Meng X, Wei T, Liu T, Wang Y, Pan Y, Wang Y. Impaired glymphatic system as evidenced by low diffusivity along perivascular spaces is associated with cerebral small vessel disease: a population-based study. Stroke Vasc Neurol. 2023 Oct;8(5):413-423. doi: 10.1136/svn-2022-002191. Epub 2023 Apr 12. PMID 37045543
- [Derived] Pan Y, Cai X, Jing J, Wang S, Meng X, Mei L, Yang Y, Jin A, DongXiao Y, Li S, Li H, Wei T, Wang Y, Wang Y. Differential associations of lipoprotein(a) level with cerebral large artery and small vessel diseases. Stroke Vasc Neurol. 2022 Jul 18;7(6):534-40. doi: 10.1136/svn-2022-001625. Online ahead of print. PMID 35851316
- [Derived] Pan Y, Jing J, Cai X, Wang Y, Wang S, Meng X, Zeng C, Shi J, Ji J, Lin J, Lyu L, Zhang Z, Mei L, Li S, Li S, Zhu W, Li H, Wei T, Wang Y. PolyvasculaR Evaluation for Cognitive Impairment and vaScular Events (PRECISE)-a population-based prospective cohort study: rationale, design and baseline participant characteristics. Stroke Vasc Neurol. 2021 Mar;6(1):145-151. doi: 10.1136/svn-2020-000411. Epub 2020 Aug 30. PMID 32863279